CLINICAL TRIAL: NCT03635632
Title: Phase I Study of Autologous T Lymphocytes Expressing GD2-specific Chimeric Antigen and Constitutively Active IL-7 Receptors for the Treatment of Patients With Relapsed or Refractory Neuroblastoma and Other GD2 Positive Solid Cancers(GAIL-N)
Brief Title: C7R-GD2.CART Cells for Patients With Relapsed or Refractory Neuroblastoma and Other GD2 Positive Cancers (GAIL-N)
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: Center for Cell and Gene Therapy, Baylor College of Medicine (Other); The Methodist Hospital Research Institute (Other); Cancer Prevention Research Institute of Texas (Other)
Responsible Party: Principal Investigator, Bilal Omer, Assistant Professor, Baylor College of Medicine
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-42207 GAIL-N
Record Dates: First submitted 2018-08-13; First posted 2018-08-17 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Relapsed Neuroblastoma; Refractory Neuroblastoma; Relapsed Osteosarcoma; Relapsed Ewing Sarcoma; Relapsed Rhabdomyosarcoma; Uveal Melanoma; Phyllodes Breast Tumor
Keywords: Gene Therapy; CAR T-cells; Neuroblastoma; chimeric antigen receptor; Immunotherapy; Sarcoma; Uveal Melanoma; Breast cancer; GD2 positive cancer
MeSH Terms: conditions — Neuroblastoma; Osteosarcoma; Sarcoma, Ewing; Rhabdomyosarcoma; Uveal Melanoma; Phyllodes Tumor; Sarcoma; Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm A: High-risk group of patients with lung metastases (Experimental): Patients will be treated at 2 dose levels without lymphodepletion chemotherapy. Three patients will be evaluated and if safety is confirmed patients will be treated at the next dose level with C7R.GD2.CART cell infusion without lymphodepletion chemotherapy.
  The protocol is divided into two arms, a high-risk group of patients with lung metastases (Arm B) and a standard risk group of all other patients (Arm A). The standard risk Arm A includes osteosarcoma patients without pulmonary disease. Each arm will undergo separate dose escalation.
  Interventions: Genetic: C7R-GD2.CART cells
- Arm B: Standard risk group of all other patients (Experimental): Patients will be treated at 2 dose levels without lymphodepletion chemotherapy. Three patients will be evaluated and if safety is confirmed patients will be treated at the next dose level with C7R.GD2.CART cell infusion without lymphodepletion chemotherapy.
  The protocol is divided into two arms, a high-risk group of patients with lung metastases (Arm B) and a standard risk group of all other patients (Arm A). The standard risk Arm A includes osteosarcoma patients without pulmonary disease. Each arm will undergo separate dose escalation.
  Interventions: Genetic: C7R-GD2.CART cells

INTERVENTIONS:
Genetic: C7R-GD2.CART cells — Active dose levels:
  C7R-GD2.CART cell without lymphodepletion (Arm A or Arm B)
  Dose Level 2b = 3 x 10^7 on day 0 and day 7
  Dose Level 3b = 1 x 10^8 on day 0 and day 7.
  Day 7 dose (+- 2 days) will be omitted if patients have persistent CRS (Grade 2 or higher) experienced a DLT or for other clinical concerns at the discretion of the PI.

SUMMARY:
This study is for patients with neuroblastoma, sarcoma, uveal melanoma, breast cancer, or another cancer that expresses a substance on the cancer cells called GD2. The cancer has either come back after treatment or did not respond to treatment. Because there is no standard treatment at this time, patients are asked to volunteer in a gene transfer research study using special immune cells called T cells. T cells are a type of white blood cell that helps the body fight infection.

The body has different ways of fighting infection and disease. No single way seems perfect for fighting cancers. This research study combines two different ways of fighting cancer: antibodies and T cells. Both antibodies and T cells have been used to treat patients with cancers. They have shown promise but have not been strong enough to cure most patients.

We have found from previous research that we can put a new gene into T cells that will make them recognize cancer cells and kill them. In our last clinical trial we made a gene called a chimeric antigen receptor (CAR) from an antibody that recognizes GD2, a substance found on almost all neuroblastoma cells (GD2-CAR). We put this gene into the patients' own T cells and gave them back to 11 neuroblastoma patients. We saw that the cells did grow for a while, but started to disappear from the blood after 2 weeks. We think that if T cells are able to last longer they may have a better chance of killing GD2 positive tumor cells.

Therefore, in this study we will add a new gene to the GD2 T cells that can cause the cells to live longer. T cells need substances called cytokines to survive and the cells may not get enough cytokines after infusion. We have added the gene C7R that gives the cells a constant supply of cytokine and helps them to survive for a longer period of time.

In other studies using T cells, investigators found that giving chemotherapy before the T cell infusion can improve the amount of time the T cells stay in the body and therefore the effect the T cells can have. This is called lymphodepletion and we think that it will allow the T cells to expand and stay longer in the body, and potentially kill cancer cells more effectively.

The GD2-C7R T cells are an investigational product not approved by the Food and Drug Administration.

The purpose of this study is to find the largest safe dose of GD2-C7R T cells, and also to evaluate how long they can be detected in the blood and what affect they have on cancer.

DETAILED DESCRIPTION:
To prepare the T cells (GD2-C7R T cells), research staff will take some blood from the patient. We will grow the GD2.C7R T cells by infecting the T cells with a retroviral vector (a special virus that can carry a new gene into cells) containing one gene that can recognize and kill cancer cells (GD2.CAR) and the new gene called C7R that will help these cells survive longer. After the new genes have been put into the T cells, the cells will be tested to make sure that they kill GD2-positive cancer cells.

Because we are growing the cells in the laboratory, we will also need to take blood to test for infectious viruses such as hepatitis and HIV (the virus that causes AIDS), and we will also ask patients to complete a questionnaire that is given to blood donors.

The cells generated will be frozen and stored to give back to the patient. Because patients will have received cells with a new gene in them patients will be followed for a total of 15 years to see if there are any long term side effects of gene transfer.

Patients will be assigned a dose of GD2-C7R T cells. The assigned dose of cells is based on body weight and height.

In this study, patients will receive the GD2-C7R cells and may also receive cyclophosphamide and fludarabine. These two drugs are standard chemotherapy medicines and may be given before the T cells to make space in the blood for the T cells to grow after receiving them.

If the patient receives cyclophosphamide and fludarabine, these drugs will be given intravenously (through an i.v. needle inserted in a vein or a central line) for 2 days and then fludarabine alone on the third day.

The patient will be given an injection of GD2-C7R T cells into the vein through an IV line at the assigned dose. Before receiving the T cell infusion, the patient may be given a dose of Benadryl (diphenhydramine) and Tylenol (acetaminophen). The infusion will take between 1 and 10 minutes. We will then monitor the patient in the clinic for about 3 hours. If you tolerate the infusion without severe side effects you may receive another infusion one week later. In this case both infusion will be considered part of one dose. The treatment will be given by the Center for Cell and Gene Therapy at Texas Children's Hospital or Houston Methodist Hospital. The patient may need to stay in Houston for up to 4 weeks after the infusion so we can monitor for side effects.

The patient will have follow-up visits after the T cell infusion at weeks 1, 2, 4, 6, and 8, then at months 3, 6, 9, and 12, and then twice a year for the next 4 years and annually for the next 10 years for a total of 15 years. The patient will also have scheduled disease evaluations after the T-cell injection at week 6 and then as clinically needed.

After disease re-evaluation, if the patient's disease has not gotten worse, or if in the future it seems the patient might benefit AND the patient has not had a severe side effect caused by the infusion of the GD2-C7R T cells, the patient may be eligible to receive one additional dose of their T cells. The dose will be at the same dose level as the first infusion and separated by at least 6 weeks such that we can make sure the patient has no severe side effects between infusions. The second dose may consist of two infusions again if you received two infusions with the first dose. If the patient receives an additional dose of GD2-C7R T-cells, then they will need to stay in Houston for up to 4 weeks after the infusion as well so we can monitor for side effects.

Medical tests before treatment--

Before being treated, the patient will receive a series of standard medical tests:

* Physical exam
* Blood tests to measure blood cells, kidney and liver function
* Measurements of the tumor by routine imaging studies and/or bone marrow evaluation. We will use the imaging studies that have been used in the past to best assess the tumor (Computer Tomogram (CT) or Magnetic Resonance Imaging (MRI), and Positron Emission Tomography (PET/CT), Bone Scan, and/or MIBG scan)
* Pulmonary Function Tests (PFT) to see how well your lungs are working

Medical tests during and after treatment--

The patient will receive standard medical tests when they are getting the infusions and afterwards:

* Physical exams
* Blood tests to measure blood cells, kidney and liver function
* Measurements of the tumor by routine imaging studies and/or bone marrow evaluation 6 weeks after the infusion (if the bone marrow showed tumor before the infusion).

To learn more about the way the GD2-C7R T cells are working and how long they last in the body, an extra amount of blood will be obtained on the day that chemotherapy starts, the day of the T-cell infusion(s) and at the end of the T-cell infusion(s), 1, 2, 4, 6 and 8 weeks after the T-cell infusion(s) and every 3 months for the 1st year, every 6 months for the next 4 years and annually for the next 10 years. The amount of blood taken will be based on weight with up to a maximum of 60 ml (12 teaspoons) of blood to be obtained at any one time. For children, the total amount of blood drawn will not be more than 3 ml (less than 1 teaspoon) per 1 kg of body weight on any one day. This volume is considered safe, but may be decreased if the patient is anemic (has a low red blood cell count).

During the time points listed above, if the GD2-C7R T cells are found in the patient's blood at a certain amount, an extra 5 ml (about 1 teaspoon) of blood may need to be collected for additional testing.

If the patient has a procedure where tumor samples are obtained, like a repeat bone marrow evaluation or tumor biopsy, we will request a sample to be used for research purposes.

The patient will receive supportive care for any acute or chronic toxicities, including blood components or antibiotics, and other intervention as appropriate.

ELIGIBILITY:
Procurement Inclusion Criteria:

1. Evaluable neuroblastoma with persistent or relapsed disease

   1. Recurrent disease following completion of aggressive multi-drug frontline therapy.
   2. Progressive disease during aggressive multi-drug frontline therapy.
   3. Primary resistant/refractory disease (less than partial response by INRC) detected at the conclusion of at least 4 cycles of aggressive multi-drug induction chemotherapy on or according to a standard high-risk treatment protocol

   OR Relapsed or refractory osteosarcoma not responsive to standard treatment

   OR Patients diagnosed with GD2 positive metastatic uveal melanoma and progressed after at least one prior systemic treatment

   OR GD2 positive breast cancer with metastatic or locally recurrent unresectable breast cancer currently progressive after at least two prior lines of therapy in the advanced setting. Patients with HER2+ disease must have failed two or more different anti-HER2 agents.

   OR Patients with other relapsed or refractory solid tumors not responsive to standard treatment with confirmed expression of GD2 by immunohistochemistry testing.
2. Life expectancy of at least 12 weeks
3. Karnofsky/Lansky score of 50% or greater
4. Absence of human anti-mouse antibodies (HAMA) prior to enrollment (only in patients that have been previously treated with murine antibodies or testing pending)
5. Informed consent and assent (as applicable) obtained from parent/guardian and child
6. Greater than 1 and less than 75 years of age

Treatment Inclusion Criteria:

1. Neuroblastoma with persistent or relapsed disease

   1. Recurrent disease following completion of aggressive multi-drug frontline therapy.
   2. Progressive disease during aggressive multi-drug frontline therapy.
   3. Primary resistant/refractory disease (less than partial response by INRC) detected at the conclusion of at least 4 cycles of aggressive multi-drug induction chemotherapy on or according to a standard high-risk treatment protocol.

   OR Relapsed or refractory osteosarcoma not responsive to standard treatment

   OR Patients diagnosed with GD2 positive metastatic uveal melanoma and progressed after at least one prior systemic treatment

   OR GD2 positive breast cancer with metastatic or locally recurrent unresectable breast cancer currently progressive after at least two prior lines of therapy in the advanced setting. Patients with HER2+ disease must have failed two or more different anti-HER2 agents.

   OR Patients with other relapsed or refractory solid tumors not responsive to standard treatment with confirmed expression of GD2 by immunohistochemistry testing.
2. Life expectancy of at least 12 weeks
3. Karnofsky/Lansky score of 50% or greater
4. Patients must have an ANC ≥ 500, platelet count ≥ 20,000
5. Pulse Ox ≥ 90% on room air
6. AST and ALT less than 5 times the upper limit of normal (less than 10 times upper normal if uveal melanoma with metastatic liver disease)
7. Total bilirubin less than 3 times the upper limit of normal
8. Serum creatinine less than 3 times upper limit of normal. Creatinine clearance is needed for patients with creatinine greater than 1.5 times upper limit of normal.
9. At least 4 weeks from completion and recovered from acute effects of all prior chemotherapy. If some effects of therapy have become chronic (i.e., treatment associated thrombocytopenia), the patient must be clinically stable and meet all other eligibility criteria. Maintenance therapy with non-investigational oral antineoplastic drugs is allowed up to 48 hours prior to infusion.
10. Absence of human anti-mouse antibodies (HAMA) prior to enrollment for patients who have received prior therapy with murine antibodies
11. Patients must have autologous activated T-cells with ≥ 20% expressing GD2.CAR
12. Informed consent and assent (as applicable) obtained from parent/guardian and child
13. Greater than 1 and less than 75 years of age

Procurement Exclusion Criteria:

1. History of hypersensitivity to murine protein containing products (patients who have undergone desensitization and successful re-challenge without hypersensitivity reaction are eligible)
2. Active autoimmune disease (requiring immunosuppressive treatment in the past 6 months)
3. Primary brain tumor or known brain metastases (on evaluation by MIBG and/or PET if applicable, CT/MRI/LP not required)

Treatment Exclusion Criteria

1. Currently receiving other investigational drugs.
2. Received any investigational immunotherapies or checkpoint inhibitors within 6 weeks. Immunotherapies include adoptive cell therapies, gene therapies, and tumor vaccines.
3. History of hypersensitivity to murine protein containing products (patients who have undergone desensitization and successful re-challenge without hypersensitivity reaction are eligible).
4. History of cardiomegaly or bilateral pulmonary infiltrates on chest radiograph or CT. However, patients with cardiomegaly on imaging may be enrolled if they have an assessment of cardiac function (i.e., ECHO or MUGA) within 3 weeks of starting protocol therapy that is within acceptable limits (LVSF>28% or LVEF>50%). Additionally, patients with bilateral pulmonary infiltrates on imaging may be enrolled if the lesions are not consistent with active neuroblastoma (i.e., negative on functional imaging with PET or MIBG, or by pathologic assessment) or not bulky in other diseases (< 5 cm for each lesion) and patient meet FiO2 criteria (>90% on room air). Baseline pulmonary function testing is required in patients with bilateral pulmonary infiltrates (except young children unable to undergo testing). Patients with poor lung function based on PFT testing (Patients with FEV 1, FVC and DLCO/diffusion capacity < 50%) will not be eligible for treatment on protocol. Patients with intermediate function (FEV 1, FVC and DLCO/diffusion capacity ≥ 50% and < 70% predicted) will require assessment by a pulmonologist prior to treatment.
5. Evidence of tumor potentially causing airway obstruction
6. Patients must not be pregnant, lactating, or unwilling to use birth control
7. Patients must not be currently receiving immunosuppressive drugs such as corticosteroids (prednisone dose of > 0.25 mg/kg/day or equivalent), tacrolimus or cyclosporine
8. Active autoimmune disease (requiring immunosuppressive treatment in the past 6 months)
9. Primary brain tumor or known brain metastases (on evaluation by MIBG and/or PET if applicable, CT/MRI/LP not required)

Ages: 1 Year to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 94 (Estimated)
Dates: Start 2019-04-23 (Actual); Primary Completion 2023-05-16 (Actual); Study Completion 2038-05-16 (Estimated)

PRIMARY OUTCOMES:
Determine maximum tolerated dose (MTD) of C7R-GD2.CART Cells | 4 weeks post T cell infusion
  Toxicity will be evaluated as per the NCI CTCAE version 5.0 with the exception of CRS and neurological toxicities that are related to T-cell infusions.

SECONDARY OUTCOMES:
Determine Anti-tumor Responses | 6 to 8 weeks post T cell infusion
  Number of patients with evaluable/measurable disease who have a partial or complete response according to standard disease evaluation criteria

CONTACTS AND LOCATIONS:
Overall Officials: Bilal Omer, MD, Principal Investigator — Baylor College of Medicine
Locations (2):
- United States (2):
  - Houston Methodist Hospital, Houston, Texas
  - Texas Children's Hospital, Houston, Texas